CLINICAL TRIAL: NCT04802980
Title: A Phase Ib, Multicenter, Open-label, Dose-escalation and Dose-expansion Study of the Safety, Tolerability and Pharmacokinetics of HB002.1T in Combination With Chemotherapy in Patients With Advanced Solid Tumors.
Brief Title: A Study of HB002.1T Plus Chemotherapy in Subjects With Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB002.1T-02
Record Dates: First submitted 2021-02-19; First posted 2021-03-17 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Paclitaxel; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HB002.1T + Oxaliplatin+ Capecitabine (Experimental): 21-24 patients with advanced gastric cancer administeredHB002.1T+ Oxaliplatin+ Capecitabine combination every 3 weeks in a 21-day cycle, total 18cycles
  Interventions: Drug: HB002.1T; Drug: Oxaliplatin; Drug: Capecitabine
- HB002.1T + Paclitaxel + Carboplatin (Experimental): 21-24 patients with advanced ovarian cancer, cervical cancer, head and neck cancer or lung cancer (not limited to the above tumor types) administered HB002.1T + Paclitaxel + Carboplatin combination every 3 weeks in a 21-day cycle, total 18cycles
  Interventions: Drug: HB002.1T; Drug: Paclitaxel; Drug: Carboplatin
- HB002.1T + Gemcitabine + Cisplatin (Experimental): 21-24 patients with advanced biliary tract tumor, pancreatic cancer, bladder cancer or nasopharyngeal carcinoma (not limited to the above tumor types) administered HB002.1T + Gemcitabine + Cisplatin combination every 3 weeks in a 21-day cycle, total 18cycles
  Interventions: Drug: HB002.1T; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: HB002.1T — HB002.1T is a vascular endothelial growth factor receptor decoy
Drug: Oxaliplatin — Oxaliplatin is an anti-tumor drug
  Arms: HB002.1T + Oxaliplatin+ Capecitabine
Drug: Capecitabine — Capecitabine is an anti-tumor drug
  Arms: HB002.1T + Oxaliplatin+ Capecitabine
Drug: Paclitaxel — Paclitaxel is an anti-tumor drug
  Arms: HB002.1T + Paclitaxel + Carboplatin
Drug: Gemcitabine — Gemcitabine is an anti-tumor drug
  Arms: HB002.1T + Gemcitabine + Cisplatin
Drug: Cisplatin — Cisplatin is an anti-tumor drug
  Arms: HB002.1T + Gemcitabine + Cisplatin
Drug: Carboplatin — Carboplatin is an anti-tumor drug
  Arms: HB002.1T + Paclitaxel + Carboplatin

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of HB002.1T in combination with different chemotherapy regimens administered to patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a Phase1b, multicenter, open-label, dose-escalation and dose-expansion in selected solid tumor indications. There are two parts to this study: a dose-escalation part and a dose-expansion part. About 63-72 subjects is planned to recruit, 27~36 subjects (9~12 subjects each arm) will be recruited during dose-escalation period The sample size may vary depending on the DLT observed at each dose level. The conventional 3+3 design will be applied for dose escalation. This trial will evaluate two adaptive dose levels, 3 to 6 subjects will be enrolled at each dose level depending on the occurrence of dose limiting toxicities (DLTs). Cohorts of 3 subjects with metastatic or locally advanced solid tumors will receive HB002.1T at escalating dose levels in combination with different chemotherapy regimens. After determination of the Maximum tolerated dose (MTD), another 12 patients in each of 3 cohorts will be added to determine the safety, tolerability, pharmacokinetic (PK), and clinical activity of HB002.1T.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤Age≤75 years
2. Histologically or cytologically confirmed advanced malignant solid tumor , including gastric cancer, ovarian cancer, cervical cancer, head and neck cancer, lung cancer, biliary tract tumor, pancreatic cancer, bladder cancer and nasopharyngeal carcinoma (not limited to the above tumor types) . And be suitable for the treatment of HB0021.T combined with 3 different chemotherapy regimen assessed by the investigators.
3. No prior radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy within 4 weeks before the first administration of HB002.1T. And no traditional herb medicines for anti-tumor within 2 weeks .
4. No prior antiangiogenic therapy such as bevacizumab, ramucirumab, apatinib or regofinib, et al.
5. At least one measurable tumor lesion as per RECIST criteria v1.1
6. ECOG performance status of 0 or 1
7. Life expectancy of at least 12 weeks
8. Meet following organ functions:

   1. Absolute neutrophil count ≥2.0 x 10^9/L(no Recombinant human granulocyte colony stimulating factor support therapy with 14 days)
   2. Hemoglobin ≥100g/L(no blood transfusion or erythropoietin support treatment was received within 14 days)
   3. Platelet count ≥100×10^9/L (No Recombinant human thrombopoietin and other supportive therapies within 14 days prior to screening phase)
   4. Serum creatinine≤1.5×ULN or creatinine clearance of≥60ml/min (based on the Cockcroft Gault formula).
   5. Serum total bilirubin≤1.5×ULN.
   6. ALT and AST ≤2.5×ULN, with the following exceptions: Patients with liver metastases assessed by investigators: AST and/or ALT≤5×ULN
   7. Blood potassium≥3.0 mmol/L, blood calcium≥2.0 mmol/L
   8. Prothrombin time (PT)≤1.2×ULN, partial prothrombin kinase time (APTT)≤1.2×ULN
   9. Urine protein < 1+showed by urine test paper, or urine protein <1g for 24 hours
9. Previous treatment toxicity returned to grade 1 as per NCI CTCAE 5.0, with the following exceptions :Hair loss or other with no safety risk judged by investigators.
10. Subjects of childbearing potential must be willing to take effective contraceptive measures throughout the study and for 3 months after the last dose of HB002.1T.And females must have a negative pregnancy test during the screening period .
11. Ability to understand the patient information and informed consent form and signed and dated written informed consent form.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  1. Confirmed active CNS metastasis and /or cancerous meningitis; For patients with stable clinical symptoms for brain metastasis for more than 3months can be enrolled.
  2. Positive test for hepatitis B, hepatitis C, or HIV at screening.
  3. History of organ transplantationHistory of severe allergy or known severe allergic reactions (greater than grade 3 in CTCAE V5.0) to macromolecular protein preparations / monoclonal antibodies and any components of the test drug;
  4. Have received other clinical trial drugs within 4 weeks before the first treatment of HB002.1T;
  5. Have undergone major surgery within 4 weeks prior to screening;
  6. Have undergone minor surgical procedures (including catheterization, except for PICC) within 2 days prior to screening;
  7. Systolic blood pressure≥140mmHg and/or diastolic blood pressure≥90mmHg after antihypertensive treatment (one antihypertensive drug is allowed in the baseline period, and the compound preparation is recognized as two);
  8. An active infection requiring antibiotics treatment during the screening period, or an unexplained fever > 38.5 °C occurs before the first dose;
  9. Hemoptysis within 4 weeks before screening (defined as coughing with ≥1 teaspoon of blood), but do not rule out cough only with sputum or small blood clot;
  10. Suffering from the following serious complications:

      1. Prior arterial thromboembolic events, venous thrombosis great than grade 3 or higher in NCI CTCAE5.0
      2. Previous or current persistent bleeding or coagulation disorders
      3. Dominant jaundice and/or coagulopathy caused by abnormal liver function
      4. Chronic Obstructive Pulmonary Disease (COPD) or other respiratory illness requiring hospitalization within 4 weeks prior to screening;
      5. History of abdominal hernia, gastrointestinal perforation abscess or acute bleeding within 6 months prior to screening;
      6. Esophageal varices, unhealed ulcer, wounds or fractures within 6 months prior to screening;
      7. Active cardiovascular diseases including but not limited to transient ischemic attack (TIA), cerebral vascular accident (CVA), transmural Myocardial infarction), transmural myocardial infarction, myocardial infarction (MI), hypertensive crisis or encephalopathy within 6 months prior to screening;
      8. Gastrointestinal disorders or conditions that may cause gastrointestinal bleeding or perforation (e.g., duodenal ulcer, intestinal obstruction, acute Crohn's disease, ulcerative colitis, massive gastrectomy and small bowel resection). Patients with chronic Crohn's disease and ulcerative colitis (except those with total colectomy and rectal resection) should be excluded even in the inactive stage
      9. Patients with hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome;
      10. Previous intestinal perforation and intestinal fistula, still not recover after surgical treatment
      11. Absorption of oral drug will be significantly affected assessed by investigators (Cohort1 only)
  11. Subjects who are in use of warfarin, heparin , aspirin (>325 mg/day) or other drugs known to inhibit platelet function within 10 days prior to the first study treatment;
  12. Subjects receiving dipyridamole, ticlopidine, clopidogrel or cilostazol treatment;
  13. Subjects with a clear history of neurological or dysfunction, such as poor adherence to epilepsy;
  14. Pregnant or nursing women;
  15. Any other reasons assessed by the investigator that are not suitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
the Maximum Tolerated Dose (MTD) of HB002.1T | up to 3 weeks
  Will be determined by dose limiting toxicity. MTD defined as the highest dose level with no more than 1 patient with DLT out of 6 patients that are treated.

SECONDARY OUTCOMES:
Immunogenicity of HB002.1T | through study completion, up to 24 weeks
  Assessed by Anti-drug Anti-body (ADA) Assay
overall response rate (ORR) | through study completion, up to 24 weeks
disease control rate (DCR) | through study completion, up to 24 weeks
Progression free survival (PFS) | through study completion, up to 24 weeks
duration of response (DOR) | through study completion, up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Ph.D, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No